CLINICAL TRIAL: NCT06216366
Title: Double-Blind, Placebo-Controlled Study Assessing the Efficacy and Safety/Tolerability of IV Rhu-pGSN as a Pre- or Post-Exposure Intervention to Mitigate Proinflammatory Responses to Decompression After High Pressure in a Hyperbaric Chamber
Brief Title: Rhu-pGSN to Mitigate Proinflammatory Responses to Decompression in Healthy SCUBA Divers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioAegis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTI-204
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Decompression Sickness
Keywords: rhu-pGSN; decompression; hyperbaric
MeSH Terms: conditions — Decompression Sickness | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Sterile normal saline 0.9% IV immediately prior to hyperbaric chamber exposure, and immediately after exposure
  Interventions: Drug: Sodium Chloride 0.9% Inj pre-exposure; Drug: Sodium Chloride 0.9% Inj post-exposure; Other: Hyperbaric chamber
- rhu-pGSN pre-exposure (Active Comparator): rhu-pGSN 24 mg/kg IV immediately prior to hyperbaric chamber exposure, and sterile normal saline 0.9% IV immediately after exposure
  Interventions: Drug: Sodium Chloride 0.9% Inj post-exposure; Drug: Recombinant human plasma gelsolin pre-exposure; Other: Hyperbaric chamber
- rhu-pGSN post-exposure (Active Comparator): Sterile normal saline 0.9% IV immediately prior to hyperbaric chamber exposure, and rhu-pGSN 24 mg/kg IV immediately after exposure
  Interventions: Drug: Sodium Chloride 0.9% Inj pre-exposure; Drug: Recombinant human plasma gelsolin post-exposure; Other: Hyperbaric chamber

INTERVENTIONS:
Drug: Sodium Chloride 0.9% Inj pre-exposure — Sterile normal saline 0.9% administered IV as a placebo immediately before hyperbaric chamber exposure
  Other Names: Normal saline
  Arms: Control; rhu-pGSN post-exposure
Drug: Sodium Chloride 0.9% Inj post-exposure — Sterile normal saline 0.9% administered IV as a placebo immediately after hyperbaric chamber exposure
  Other Names: Normal saline
  Arms: Control; rhu-pGSN pre-exposure
Drug: Recombinant human plasma gelsolin pre-exposure — rhu-pGSN administered IV at a dose of 24 mg/kg immediately before hyperbaric chamber exposure
  Other Names: rhu-pGSN
  Arms: rhu-pGSN pre-exposure
Drug: Recombinant human plasma gelsolin post-exposure — rhu-pGSN administered IV at a dose of 24 mg/kg immediately after hyperbaric chamber exposure
  Other Names: rhu-pGSN
  Arms: rhu-pGSN post-exposure
Other: Hyperbaric chamber — High-pressure profile equivalent 35 minutes at a depth of 30 meters of sea water

SUMMARY:
Healthy trained SCUBA divers will be randomized into three groups and exposed to a high-pressure profile in a hyperbaric chamber. The high-pressure profile simulates the pressure at a depth of 30 meters of sea water (MSW) for 35 minutes. In the control group, the subjects will receive intravenous normal saline immediately before and after the high-pressure exposure. The second group will receive intravenous recombinant human gelsolin (rhu-pGSN) 24 mg/kg immediately prior to the exposure, and saline post-exposure. The third group will receive saline pre-exposure and rhu-pGSN post-exposure. Blood samples will be collected at multiple time points pre- and post-exposure to assess levels of inflammatory markers, including interleukin (IL)-1β. Other assessments include screening for gas bubbles, a validated questionnaire to assess the incidence of clinical decompression sickness (DCS), measurement of plasma gelsolin (pGSN) levels, and measurement of anti-pGSN antibodies.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study in healthy volunteers who have been trained for SCUBA diving.

The study will be performed in the hyperbaric chamber at the University of Maryland. Healthy trained divers will be exposed to a high-pressure profile known to cause decreased plasma gelsolin (pGSN), increased microparticles (MPs), and cytokine changes with no adverse effects such as decompression sickness (DCS). The intervention with recombinant human plasma gelsolin (rhu-pGSN) is patterned after the animal model of DCS where rhu-pGSN administration prior to or after decompression abrogated organ injuries concurrent with inhibiting elevations of MPs and intra-particle interleukin (IL)-1β concentration.

There will be three experimental groups. The control subjects will receive intravenous sterile 0.9% saline immediately before and immediately after the 35-minute 30 meters of sea water (MSW) exposure. A second group will receive intravenous rhu-pGSN 24 mg/kg immediately prior to the high pressure exposure and sterile saline post-exposure. The third group will receive sterile saline prior to the exposure and 24 mg/kg rhu-pGSN post-exposure. Development of DCS is not anticipated based on previous experience with 30 MSW exposure for 35 minutes.

Once informed consent is obtained, the following assessments/procedures will be performed:

1. Confirm the potential participant is healthy and has been trained as a SCUBA diver.
2. Record medical history, including concomitant medications.
3. Perform pregnancy test (urine or blood) for women of childbearing potential.
4. Perform vital signs and physical examination.
5. Perform EKG.
6. Measure CBC and metabolic profile lab tests at local laboratory.
7. Collect pretreatment blood samples for measurement of pGSN and analysis of antibodies against pGSN.
8. Perform Cardiac Echo for bubbles.
9. Collect aliquots of blood for subsequent biomarker assays (including IL-1β, pGSN, nitric oxide synthase [NOS2], tumor necrosis factor [TNF]) and microparticles for analysis.
10. If eligibility criteria are satisfied, the subject will be randomized 1:1:1 (rhu-pGSN pre high pressure exposure:rhu-pGSN post high pressure exposure:saline placebo). After reconstitution to 200 mg in a final volume of 5 mL in a 10-mL vial, rhu pGSN is not to be kept at room temperature for >2 hours prior to beginning the IV push. Study drug is administered by an IV push through a 0.2 μm filter. The syringe, filter, and extension tubing for the IV push of study drug are to be connected as close to the subjects as possible. Each subject will receive 2 IV study injections. No subject will receive more than 1 dose of rhu-pGSN.
11. Subject will be exposed to high pressure (30 meters salt water [MSW] for 35 minutes) and followed up for 24 hours and again at day 14.
12. A well-being questionnaire will be administered.

Before the 30 MSW exposure, blood will be obtained from all subjects for pre-exposure measurements. A second sampling will be obtained after 30 minutes post initiation of the exposure to high pressure while still at pressure in the hyperbaric chamber and before decompression to assess whether inflammatory changes occurring due to pressure and before decompression are altered by rhu-pGSN when administered pre-exposure to high pressure. Blood specimens will be obtained at 60, 120 and 240 minutes after decompression.

Prior to, and following the 30 MSW exposure, all subjects will be screened for gas bubbles (vascular gas emboli [VGE]) using a phase array ultrasonic probe. Intravascular bubbles are thought to play a role in the evolution of DCS. Preliminary work has demonstrated that rhu-pGSN can lyse inflammatory MPs and ~28% of MPs contain a gas phase of nitrogen dioxide that can serve as a nucleation site for bubble formation. Therefore, this work will also evaluate whether rhu-pGSN can prevent bubble production.

The Doolette well-being questionnaire will be administered 60 minutes after decompression.

On Day 14 blood samples for analysis of antibodies against pGSN are to be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Experienced healthy trained female or male SCUBA divers without known underlying comorbidities
2. Age ≥18
3. Informed consent obtained from subject
4. During the course of the study starting at screening and for at least 3 months after their final study treatment:

   * Female subjects of childbearing potential must agree to use 2 medically accepted and approved birth control methods
   * Male subjects with a partner who might become pregnant must agree to use reliable forms of contraception (i.e., vasectomy, abstinence), or an acceptable method of birth control must be used by the partner
   * All subjects must agree not to donate sperm or eggs

Exclusion Criteria:

1. Any co-morbidity contraindicating SCUBA diving
2. Pregnant or lactating women
3. History of unrepaired cardiac shunt or echocardiographic evidence of patent foramen ovale or atrial septal defect
4. Any active underlying conditions including but not limited to cancer or other illness treated with systemic chemotherapy, immunomodulatory biologics, or radiation therapy during the last 360 days or expected to be treated in the upcoming 120 days
5. Refusal or inability to use adequate contraception
6. Participation in an investigational clinical trial (e.g., device, drug, or biologic) in the previous 30 days
7. Any acute illness or vaccination in the previous 30 days
8. History of alcohol or recreation drug use disorder
9. Known allergy to study drug or excipients
10. Weight >125 kg
11. Unsuitable for study participation, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Interleukin (IL)-1β | At baseline, during and after exposure, and afterward at 60, 120, and 240 minutes, at 24 hours, and at day 14
  Change from baseline in blood IL-1β levels at 2 hours after hyperbaric chamber exposure
Adverse Events | 14 days
  Incidence, causality, and severity of Adverse Events (graded according to the NCI CTCAE version 5.0)

SECONDARY OUTCOMES:
Biomarkers | At baseline, during and after exposure, and afterward at 60, 120, and 240 minutes, at 24 hours, and at day 14
  Change from baseline in biomarker levels, including but not limited to: NOS2, TNFα, IL-6, CCL2, CCL5, and microparticles
Gas bubbles | At baseline, and 30, 60, 120, and 240 minutes after exposure
  Cardiac Echo to screen for vascular gas emboli (VGE) using a phase array ultrasonic probe
Questionnaire | 60 minutes after hyperbaric chamber exposure
  Doolette well-being questionnaire to screen for clinical decompression sickness (DCS)
pGSN levels | At baseline, during and after exposure, and afterward at 240 minutes, at 24 hours, and at day 14
  Blood levels of plasma gelsolin
anti-pGSN antibodies | Baseline, and at day 14
  Blood levels of anti-plasma gelsolin antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No